CLINICAL TRIAL: NCT04876573
Title: Pilot Study for Cyproheptadine in Hospitalized Patient for COVID-19: a Single-center, Observational Retrospective-prospective Comparative Study.
Brief Title: Pilot Study for Cyproheptadine in Hospitalized Patient for COVID-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-2669
Record Dates: First submitted 2021-05-03; First posted 2021-05-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: Viral Pneumonia; COVID-19 Pneumonia; Serotonin Syndrome; Platelet Dysfunction
MeSH Terms: conditions — Pneumonia, Viral; Serotonin Syndrome | interventions — Cyproheptadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cyproheptadine (Experimental)
  Interventions: Drug: Cyproheptadine Hydrochloride 4 MG

INTERVENTIONS:
Drug: Cyproheptadine Hydrochloride 4 MG — Phase 1: Cyproheptadine 4 mg three time a day for 10 days, per oral administration associated to Standard care of COVID 19 patient currently recommend by WHO
  Phase 2: Cyproheptadine 8 mg three time a day for 10 days, per oral administration associated to Standard care of COVID 19 patient currently recommend by WHO
  The dose will be adjusted according to the renal function.

SUMMARY:
This is a Pilot study for evaluating the feasibility, security and efficacy of the use of Cypropheptadine, an antihistaminic and antiserotonin drug, as an adjunct of the standardized treatment in a population of patient who are hospitalized and requiring oxygen therapy for COVID-19.

DETAILED DESCRIPTION:
Background :

Biochemical studies have revealed a significant increase in plasma serotonin levels in patients suffering from COVID-19 multi-organ disease, which appears to be a consequence of platelet hyperreactivity and dysfunction.

Among the several potential therapeutic pathways available to modulate this serotonin dysregulation is the use of cyproheptadine, an Anti-serotonergic antihistamine that can potentially improve organ dysfunction related to elevated plasma serotonin levels.

The investigators hypothesize that treatment with cyproheptadine will improve clinical course in these patients.

Objectives:

Primary objective

Compare the clinical course according to the WHO ordinal severity score for COVID-19, between a retrospective and a prospective interventional cohort of patient hospitalized in the same hospital.

Secondary objectives

Evaluate the safety of the use of the cyproheptadine hospitalized patients presenting COVID 19.

Evaluate the study in term of Feasibility Recruitment rate and Study completion rate.

Evaluate the outcome in term of Death, Needs of Non-invasive and/or invasive mechanical ventilation and Total Length of hospitalization Evaluate the evolution of clinical indicators of oxygenation and blood parameters of inflammation, renal function, hepatic cytolysis and platelet count.

Design:

This pilot trial is a non-blinded clinical designed to access the feasibility, the security and the efficacy of the use of Cyproheptadine in patient hospitalized in a single center for Covid-19 with comparison between:

A retrospective cohort study of patient and treated by standard care according to WHO international guidelines.

A prospective study of a cohort of patients hospitalized for covid 19 taking oral Cyproheptadine during 10 days in addition to standard care according to WHO international guidelines. The prospective study will be divided into two different phases in which two different doses of cyproheptadine will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Women and men aged 18 and over.
* Requiring treatment for COVID 19 and whose clinical status corresponds to a score equal to or greater than 5 on the WHO Clinical Progression Scale.
* For the prospective study, able to give informed consent.
* Not presenting an exclusion criterion

Exclusion Criteria:

* Pregnancy
* Patients with pre-existing terminal condition with life expectancy < 6 months
* Patient with clinically frailty according to a score of the clinical frailty scale equal or superior to 7
* Patients with pre-existing severe lung disease requiring home oxygen therapy.
* Patients with pre-existing severe hepatic cirrhosis (Grade C according to the Child-Pugh classification)
* Patients with pre-existing kidney failure (GFR strictly less than 15ml/min/1.73m2 according The KDIGO classification) or requiring renal replacement therapy.
* Patients with pre-existing angle-closure glaucoma
* Patient with symptomatic prostatic hypertrophy or bladder neck obstruction
* Patient with history of seizure disorder
* Patient with history of adverse reaction to antihistamines or to Cyproheptadine
* Patients taking routinely SSRI or monoamine oxidase inhibitor therapy.
* Patients presenting severe hepatic cytolysis with ALP >5 ULN at the time of study inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Clinical evolution according the WHO Clinical Progression Scale | Approximately 28 days
  World Health Organisation Clinical Progression Scale for COVID 19 Minimal value 0 (uninfected) to maximal value 10 (Dead)

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Approximately 28 days
  Safety evaluation, as measured by suspected as related to cyproheptadine during the first 28 days after inclusion in the study:
  Adverse events
  Adverse drug reactions
  Serious adverse event and adverse drug reaction
Recruitement rate | 6 month
Completion rate | 6 month
Rate of Death from any cause | Approximately 28 days
Total number of days of hospitalisation | Approximately 28 days
Total number of days of hospitalization in the ICU | Approximately 28 days
Total number of days of mechanical ventilation | Approximately 28 days
Daily ROX ratio | Approximately 28 days
  Worst value of ROX ratio (SPO2/FiO2/Respiratory Rate) at D3,5,7,10,14,28
Creatinine level | Approximately 28 days
  Worst value of Laboratory assessment of Creatinine at Days 3,5,7,10,14,28 after inclusion in the study
Alanine amino transferase level | Approximately 28 days
  Worst value of Laboratory assessment of Alanine amino transferase at Days 3,5,7,10,14,28 after inclusion in the study
C Reactive Protein level | Approximately 28 days
  Worst value of Laboratory assessment of CRP at Days 3,5,7,10,14,28 after inclusion in the study
D-Dimere level | Approximately 28 days
  Worst value of Laboratory assessment of D-Dimere at Days 3,5,7,10,14,28 after inclusion in the study
Platelet count | Approximately 28 days
  Worst value of Laboratory assessment of platelet count at Days 3,5,7,10,14,28 after inclusion in the study